CLINICAL TRIAL: NCT00091572
Title: Extended Schedule, Escalated Dose Temozolomide Versus Dacarbazine in Stage IV Metastatic Melanoma: A Randomized Phase III Study of the EORTC Melanoma Group
Brief Title: Temozolomide Versus Dacarbazine in Stage IV Metastatic Melanoma (Study P03267)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P03267; NCT00101218 (obsolete NCT alias)
Record Dates: First submitted 2004-09-10; First posted 2004-09-14 (Estimated); Results first posted 2009-03-12 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-05

CONDITIONS: Melanoma
Keywords: Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — Temozolomide; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): temozolomide 150 mg/m2/day PO, on 7 consecutive days every 14 days ("7 days on / 7 days off" continuously)
  Interventions: Drug: Temozolomide
- B (Active Comparator): dacarbazine 1000 mg/m2 IV, on Day 1 +/- 3 days every 3 weeks
  Interventions: Drug: Dacarbazine

INTERVENTIONS:
Drug: Temozolomide — oral capsule; 150 mg/m2/day PO (by mouth), on 7 consecutive days every 14 days ("7 days on / 7 days off" continuously); one cycle of temozolomide is defined as a 6-week period; treatment will continue until progression of the disease, unacceptable toxicity, subject refusal, or opinion of the treating physician that it is in the subject's best interest to stop.
  Other Names: Temodal, Temodar, SCH 52365
  Arms: A
Drug: Dacarbazine — intravenous solution; dacarbazine 1000 mg/m2 IV (in the vein), on Day 1 +/- 3 days every 3 weeks; one cycle of dacarbazine is defined as a 3-week period; treatment will continue until progression of the disease, unacceptable toxicity, subject refusal, or opinion of the treating physician that it is in the subject's best interest to stop.
  Other Names: DTIC-Dome
  Arms: B

SUMMARY:
The purpose of this study is to ascertain if the extended schedule of Temozolomide, which allows increased doses and potential depletion of the enzyme underlaying resistance, is a more effective treatment of metastatic melanoma than single agent dacarbazine.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, stage IV, surgically incurable melanoma
* Age 18 years or older
* World Health Organization (WHO) Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Meets protocol requirements for specified laboratory values
* Must be able to take oral medication
* Must be disease free from cancer for period of 5 years (except for surgically cured carcinoma in-situ of the cervix and basal or squamous cell carcinoma of the skin).
* Women of childbearing potential and men must be practicing a medically approved contraception.
* Must provide written informed-consent to participate in the study.
* Must have full recovery from major surgery or adjuvant treatment
* No clinically uncontrolled infectious disease including HIV or AIDS-related illness

Exclusion Criteria:

* Ocular melanomas
* Brain Metastases
* Prior cytokine or chemotherapy for stage IV disease
* Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 859 (Actual)
Dates: Start 2004-10-20 (Actual); Primary Completion 2007-12-31 (Actual); Study Completion 2007-12-31 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Patel PM, Suciu S, Mortier L, Kruit WH, Robert C, Schadendorf D, Trefzer U, Punt CJ, Dummer R, Davidson N, Becker J, Conry R, Thompson JA, Hwu WJ, Engelen K, Agarwala SS, Keilholz U, Eggermont AM, Spatz A; EORTC Melanoma Group. Extended schedule, escalated dose temozolomide versus dacarbazine in stage IV melanoma: final results of a randomised phase III study (EORTC 18032). Eur J Cancer. 2011 Jul;47(10):1476-83. doi: 10.1016/j.ejca.2011.04.030. Epub 2011 May 18. PMID 21600759

RESULTS

PARTICIPANT FLOW:
Groups:
- Temozolomide: temozolomide 150 mg/m2/day PO, on 7 consecutive days every 14 days ("7 days on / 7 days off" continuously)
- Dacarbazine: dacarbazine 1000 mg/m2 IV, on Day 1 +/- 3 days every 3 weeks
Period: Overall Study
Arm/Group | Temozolomide | Dacarbazine
Started | 429 (10 subjects in temozolomide group not treated.) | 430 (9 subjects in dacarbazine group not treated.)
Completed | 334 (Progressive disease/relapse/death due to progressive disease) | 348 (Progressive disease/relapse/death due to progressive disease)
Not Completed | 95 | 82
Not completed — Lost to Follow-up | 1 | 1
Not completed — Subject's Refusal unrelated to toxicity | 14 | 22
Not completed — Death not due to malignancy/toxicity | 1 | 3
Not completed — Medical Decision unrelated toxicity/PD | 10 | 22
Not completed — Other Reason | 6 | 13
Not completed — Ongoing (still on treatment) | 8 | 12
Not completed — Major Protocol Violation | 2 | 0
Not completed — Toxicity (Related AE) | 53 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Temozolomide | Dacarbazine | Total
Number analyzed (Participants) | 429 | 430 | 859
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 276 | 261 | 537
  >=65 years | 153 | 169 | 322
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 179 | 177 | 356
  Male | 250 | 253 | 503

OUTCOME MEASURES:

1. Secondary Outcome: Progression Free Survival
Description: Progression free survival was defined as the time from the date of randomization to the date of disease progression or the date of death regardless of the cause.
Time Frame: Treatment continued until disease progression or unacceptable toxicity. Patients will be followed for survival.
Population: Intent to Treat Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Temozolomide | Dacarbazine
Number analyzed (Participants) | 429 | 430
Months | 2.30 [2.23 to 2.43] | 2.17 [2.14 to 2.27]
Statistical Analysis 1: Comparison: Temozolomide vs Dacarbazine; Test type: Superiority or Other; p = 0.2663, Log Rank; Hazard Ratio (HR) = 0.92, 95% CI [0.80 to 1.06] — Temozolomide events (progressions/deaths) = 401. Dacarbazine events (progressions/deaths) = 398

2. Primary Outcome: Overall Survival
Description: Overall Survival was defined as the time from the date of randomization to the date of death from any cause.
Time Frame: The final analysis was to be performed when at least 616 deaths had occurred.
Population: Intent to Treat Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Temozolomide | Dacarbazine
Number analyzed (Participants) | 429 | 430
Months | 9.13 [8.11 to 9.89] | 9.36 [8.21 to 10.28]
Statistical Analysis 1: Comparison: Temozolomide vs Dacarbazine; Test type: Superiority or Other; p = 0.9999, Log Rank; Hazard Ratio (HR) = 1.00, 95% CI [0.86 to 1.17] — Temozolomide events (deaths) = 320. Dacarbazine events (deaths) = 325

3. Secondary Outcome: Objective Response Rate in Subjects With Measurable Lesions
Description: Based on investigator's assessment of response in subjects with measurable lesions. Objective response = complete response + partial response. Complete response = disappearance of all target lesions. Partial response = at least a 30% decrease in the sum of longest diameter of target lesions taking as reference the baseline sum longest diameter.
Time Frame: Treatment continued until disease progression or unacceptable toxicity.
Population: Intent to treat population with measurable disease at Baseline.
Measure: Median (95% Confidence Interval); unit: Ratio
Arm/Group | Temozolomide | Dacarbazine
Number analyzed (Participants) | 401 | 388
Ratio | 0.14 [0.10 to 0.17] | 0.10 [0.07 to 0.12]
Statistical Analysis 1: Comparison: Temozolomide vs Dacarbazine; Test type: Superiority or Other; p = 0.0718, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.43, 95% CI [0.97 to 2.12] — Temozolomide numerator (responders) = 55. Dacarbazine numerator (responders) = 37

4. Secondary Outcome: Duration of Objective Response
Description: Duration of objective response was measured from the time the criteria were met for complete response or partial response to the first date that recurrent or progressive disease was objectively documented.
Time Frame: Treatment continued until disease progression or unacceptable toxicity.
Population: All responders
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Temozolomide | Dacarbazine
Number analyzed (Participants) | 55 | 37
Months | 4.34 [4.17 to 6.18] | 8.31 [6.08 to 19.25]

ADVERSE EVENTS:
Arm/Group | Temozolomide | Dacarbazine
Serious Adverse Events (participants affected / at risk) | 124/419 | 100/421
Other Adverse Events (participants affected / at risk) | 394/419 | 374/421
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide (N=419) | Dacarbazine (N=421)
ANAEMIA HAEMOLYTIC AUTOIMMUNE (Blood and lymphatic system disorders) | 2 (6) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
NORMOCHROMIC NORMOCYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 (1) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 1 (1) | 0 (0)
ARRHYTHMIA SUPRAVENTRICULAR (Cardiac disorders) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 3 (3) | 1 (2)
ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 0 (0) | 1 (1)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 (1) | 1 (1)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 (0) | 1 (1)
NODAL ARRHYTHMIA (Cardiac disorders) | 0 (0) | 1 (1)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (1) | 1 (1)
SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0 (0) | 1 (1)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
GLAUCOMA (Eye disorders) | 0 (0) | 1 (1)
KERATITIS (Eye disorders) | 1 (1) | 0 (0)
PHOTOPHOBIA (Eye disorders) | 1 (1) | 0 (0)
UVEITIS (Eye disorders) | 0 (0) | 1 (1)
VISION BLURRED (Eye disorders) | 1 (1) | 0 (0)
VITREOUS HAEMORRHAGE (Eye disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 6 (9) | 8 (8)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 1 (1)
ASCITES (Gastrointestinal disorders) | 0 (0) | 1 (3)
COLONIC FISTULA (Gastrointestinal disorders) | 0 (0) | 1 (1)
COLONIC OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 6 (10) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 4 (4)
HAEMATEMESIS (Gastrointestinal disorders) | 2 (2) | 0 (0)
INTRA-ABDOMINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 11 (14) | 10 (12)
PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
SMALL INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 1 (1)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 15 (21) | 9 (11)
CHEST PAIN (General disorders) | 1 (2) | 2 (2)
CHILLS (General disorders) | 1 (1) | 2 (3)
FATIGUE (General disorders) | 7 (9) | 5 (6)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 4 (4) | 3 (3)
MULTI-ORGAN FAILURE (General disorders) | 1 (1) | 1 (1)
PERFORMANCE STATUS DECREASED (General disorders) | 1 (1) | 1 (2)
PYREXIA (General disorders) | 3 (3) | 8 (9)
CHOLANGITIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (2) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (2) | 0 (0)
HEPATIC FAILURE (Hepatobiliary disorders) | 1 (2) | 0 (0)
HEPATIC PAIN (Hepatobiliary disorders) | 1 (1) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 2 (2)
ABSCESS INTESTINAL (Infections and infestations) | 1 (1) | 1 (1)
APPENDICITIS (Infections and infestations) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0)
CYSTITIS (Infections and infestations) | 0 (0) | 1 (1)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 2 (2)
ENDOCARDITIS (Infections and infestations) | 1 (1) | 0 (0)
ERYSIPELAS (Infections and infestations) | 0 (0) | 1 (1)
GASTROINTESTINAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
HAEMOPHILUS INFECTION (Infections and infestations) | 0 (0) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 1 (1) | 0 (0)
INFECTION (Infections and infestations) | 1 (1) | 1 (1)
INFECTIVE MYOSITIS (Infections and infestations) | 0 (0) | 1 (1)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
LUNG INFECTION (Infections and infestations) | 0 (0) | 2 (3)
PNEUMONIA (Infections and infestations) | 4 (4) | 1 (1)
RHINITIS (Infections and infestations) | 1 (2) | 0 (0)
SALPINGITIS (Infections and infestations) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 4 (4) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 1 (1) | 0 (0)
SERRATIA INFECTION (Infections and infestations) | 1 (1) | 0 (0)
SKIN INFECTION (Infections and infestations) | 0 (0) | 1 (1)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
TOOTH ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 2 (2)
WOUND INFECTION (Infections and infestations) | 2 (3) | 1 (1)
AORTIC INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (3) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 1 (3)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 1 (3)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (1) | 1 (1)
BLOOD CALCIUM INCREASED (Investigations) | 1 (1) | 0 (0)
BLOOD GLUCOSE DECREASED (Investigations) | 0 (0) | 2 (2)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 2 (6) | 0 (0)
BLOOD POTASSIUM DECREASED (Investigations) | 1 (1) | 0 (0)
HAEMOGLOBIN DECREASED (Investigations) | 3 (5) | 7 (9)
LYMPHOCYTE COUNT DECREASED (Investigations) | 3 (5) | 0 (0)
MINI MENTAL STATUS EXAMINATION ABNORMAL (Investigations) | 0 (0) | 1 (1)
NEUTROPHIL COUNT DECREASED (Investigations) | 9 (14) | 3 (4)
PLATELET COUNT DECREASED (Investigations) | 21 (34) | 3 (4)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 5 (7) | 2 (4)
ANOREXIA (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (6)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
OSTEOLYSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
SOFT TISSUE NECROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
ATAXIA (Nervous system disorders) | 3 (3) | 1 (1)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 0 (0)
COGNITIVE DISORDER (Nervous system disorders) | 1 (1) | 0 (0)
CONUS MEDULLARIS SYNDROME (Nervous system disorders) | 1 (1) | 0 (0)
CONVULSION (Nervous system disorders) | 2 (2) | 2 (2)
DIZZINESS (Nervous system disorders) | 3 (5) | 2 (3)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 1 (1) | 2 (2)
HEADACHE (Nervous system disorders) | 5 (5) | 2 (2)
HEMIPLEGIA (Nervous system disorders) | 0 (0) | 1 (1)
INTRACRANIAL PRESSURE INCREASED (Nervous system disorders) | 0 (0) | 1 (1)
MEMORY IMPAIRMENT (Nervous system disorders) | 0 (0) | 1 (1)
NEURALGIA (Nervous system disorders) | 1 (1) | 1 (1)
NEUROLOGICAL SYMPTOM (Nervous system disorders) | 0 (0) | 1 (1)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 (0) | 2 (2)
SOMNOLENCE (Nervous system disorders) | 1 (1) | 1 (1)
SPINAL CORD COMPRESSION (Nervous system disorders) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
SYNCOPE VASOVAGAL (Nervous system disorders) | 0 (0) | 2 (2)
ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1) | 2 (2)
DEPRESSION (Psychiatric disorders) | 2 (2) | 1 (1)
DRUG DEPENDENCE (Psychiatric disorders) | 0 (0) | 1 (1)
HAEMORRHAGE URINARY TRACT (Renal and urinary disorders) | 0 (0) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 2 (5) | 0 (0)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 (2) | 0 (0)
URETERIC OBSTRUCTION (Renal and urinary disorders) | 3 (5) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 1 (1)
MENORRHAGIA (Reproductive system and breast disorders) | 1 (2) | 0 (0)
PELVIC PAIN (Reproductive system and breast disorders) | 1 (1) | 0 (0)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 4 (5)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
PLEURAL FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
EXFOLIATIVE RASH (Skin and subcutaneous tissue disorders) | 5 (12) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ABDOMINAL CAVITY DRAINAGE (Surgical and medical procedures) | 1 (3) | 0 (0)
LYMPHADENECTOMY (Surgical and medical procedures) | 2 (2) | 1 (1)
MALIGNANT TUMOUR EXCISION (Surgical and medical procedures) | 2 (3) | 0 (0)
MASTECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0)
PLEURODESIS (Surgical and medical procedures) | 1 (1) | 0 (0)
SKIN LESION EXCISION (Surgical and medical procedures) | 1 (2) | 1 (1)
THORACIC CAVITY DRAINAGE (Surgical and medical procedures) | 1 (1) | 0 (0)
HAEMATOMA (Vascular disorders) | 1 (4) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 2 (2)
HYPOTENSION (Vascular disorders) | 1 (1) | 3 (4)
THROMBOSIS (Vascular disorders) | 1 (2) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide (N=419) | Dacarbazine (N=421)
ABDOMINAL PAIN (Gastrointestinal disorders) | 43 (91) | 31 (58)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 22 (43) | 17 (33)
CONSTIPATION (Gastrointestinal disorders) | 183 (563) | 111 (267)
DIARRHOEA (Gastrointestinal disorders) | 79 (146) | 71 (139)
DYSPEPSIA (Gastrointestinal disorders) | 22 (85) | 25 (47)
NAUSEA (Gastrointestinal disorders) | 286 (966) | 206 (535)
VOMITING (Gastrointestinal disorders) | 211 (456) | 103 (208)
FATIGUE (General disorders) | 253 (1102) | 240 (798)
INFLUENZA LIKE ILLNESS (General disorders) | 18 (30) | 24 (37)
OEDEMA PERIPHERAL (General disorders) | 30 (90) | 37 (136)
PYREXIA (General disorders) | 49 (67) | 54 (71)
WEIGHT DECREASED (Investigations) | 87 (380) | 45 (114)
WEIGHT INCREASED (Investigations) | 16 (90) | 40 (209)
ANOREXIA (Metabolism and nutrition disorders) | 118 (384) | 79 (157)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 20 (66) | 23 (79)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 35 (88) | 47 (102)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 35 (120) | 31 (54)
DIZZINESS (Nervous system disorders) | 51 (135) | 45 (77)
DYSGEUSIA (Nervous system disorders) | 22 (77) | 17 (35)
HEADACHE (Nervous system disorders) | 92 (206) | 56 (115)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 28 (75) | 29 (77)
DEPRESSION (Psychiatric disorders) | 25 (81) | 19 (49)
INSOMNIA (Psychiatric disorders) | 25 (66) | 17 (42)
COUGH (Respiratory, thoracic and mediastinal disorders) | 71 (193) | 51 (91)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 45 (109) | 48 (105)
EXFOLIATIVE RASH (Skin and subcutaneous tissue disorders) | 51 (156) | 23 (45)
PRURITUS (Skin and subcutaneous tissue disorders) | 75 (214) | 29 (67)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other